CLINICAL TRIAL: NCT05312398
Title: CAPRI 2 GOIM Study: Investigate the Efficacy and Safety of a Bio- Marker-driven Cetuximab-based Treatment Regimen Over 3 Treatment Lines in mCRC Patients With RAS/BRAF wt Tumors at Start of First Line
Brief Title: CAPRI 2 GOIM Study: Investigate the Efficacy and Safety of a Bio-marker Driven Cetuximab-based Treatment Regimen
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Fortunato Ciardiello, Principal Investigator, University of Campania Luigi Vanvitelli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPRI2-MS062202-0123
Record Dates: First submitted 2022-03-01; First posted 2022-04-05 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Adenocarcinoma
MeSH Terms: interventions — Cetuximab; IFL protocol; Folfox protocol; Irinotecan

STUDY DESIGN:
Intervention Model Description: 3 treatment lines in mCRC patients with RAS/BRAF wt tumors at start of first line.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): This is an open-label phase II study investigating the efficacy and safety of a bio-marker-driven cetuximab-based treatment regimen over 3 treatment lines in mCRC patients with RAS/BRAF wt tumors at start of first line. Based on dynamic and longitudinal liquid biopsy assessment of RAS/BRAF status, that will be prospectively performed before each line of treatment, mCRC patients will be treated with cetuximab in combination with chemotherapy throughout three lines of therapy, as follows:
  * FOLFIRI plus cetuximab (first line);
  * FOLFOX plus cetuximab (second line);
  * irinotecan plus cetuximab (third line).
  If at progression after the first line or after the second line, the liquid biopsy assessment indicates RAS and or BRAF mutant status, patients will be treated with FOLFOX plus bevacizumab as second line of therapy, or with regorafenib or with trifluridine-tipiracil (investigator's choice) as third line therapy.
  Interventions: Drug: Cetuximab; Drug: FOLFIRI; Drug: FOLFOX regimen; Drug: Irinotecan

INTERVENTIONS:
Drug: Cetuximab — I LINE:
  - FOLFIRI + cetuximab
  FOLFIRI: 200 mg L-folinic acid with 180 mg/ m² irinotecan over 1.30 h IV infusion, followed by a 400 mg/ m² IV bolus of fluorouracil followed by 2400 mg/ m² fluorouracil IV infusion over 46 h every 14 days.
  Cetuximab: 400 mg/m2 initial dose (120-minute IV infusion on cycle 1 day 1), then 250 mg/m2 once weekly thereafter
  II LINE:
  - FOLFOX + cetuximab
  FOLFOX: 200 mg L-folinic acid given concurrently with 85 mg/ m² oxaliplatin over 2 h IV infusion, followed by a 400 mg/ m² IV bolus of fluorouracil followed by 2400 mg/ m² fluorouracil IV infusion over 46 h every 14 days.
  Cetuximab: as I line
  THIRD LINE:
  - Irinotecan + cetuximab
  Irinotecan: 180 mg/ m² irinotecan over 1.30 h, IV infusion every 2 weeks. Cetuximab: as I line
  Other Names: Erbitux
Drug: FOLFIRI — I LINE:
  - FOLFIRI + cetuximab
  FOLFIRI: 200 mg L-folinic acid given concurrently with 180 mg/ m² irinotecan over 1.30 h IV infusion, followed by a 400 mg/ m² IV bolus of fluorouracil followed by 2400 mg/ m² fluorouracil IV infusion over 46 h every 14 days.
  Cetuximab: 400 mg/m2 initial dose (120-minute IV infusion on cycle 1 day 1), then 250 mg/m2 once weekly thereafter
Drug: FOLFOX regimen — II LINE:
  - FOLFOX + cetuximab
  FOLFOX: 200 mg L-folinic acid given concurrently with 85 mg/ m² oxaliplatin over 2 h IV infusion, followed by a 400 mg/ m² IV bolus of fluorouracil followed by 2400 mg/ m² fluorouracil IV infusion over 46 h every 14 days.
  Cetuximab: as I line
  Other Names: FOLFOX
Drug: Irinotecan — III LINE:
  - Irinotecan + cetuximab
  Irinotecan: 180 mg/ m² irinotecan over 1.30 h, IV infusion every 2 weeks. Cetuximab: as I line

SUMMARY:
This clinical program aims to evaluate the activity and efficacy of cetuximab continuation of treatment for three lines of therapy with rotation of chemotherapy (FOLFIRI, FOLFOX, irinotecan) in mCRC patients, whose tumors remain RAS/BRAF WT. The study will also evaluate the activity and efficacy of cetuximab re-introduction in combination with irinotecan as third line therapy in the concept of re-challenge for those patients that will be treated in second line with chemotherapy plus anti-angiogenic drugs (FOLFOX plus bevacizumab), having a RAS or BRAF mutant disease at the time of progression after FOLFIRI plus cetuximab first line treatment. A novel characteristic of this program is that the therapeutic algorithm will be defined at each treatment decision (first line, second line and third line) in a prospective fashion in each patient by liquid biopsy assessment of RAS/BRAF status.

DETAILED DESCRIPTION:
Based on dynamic and longitudinal liquid biopsy assessment of RAS/BRAF status, that will be prospectively performed before each line of treatment, mCRC patients will be treated with cetuximab in combination with chemotherapy throughout three lines of therapy, as follows: FOLFIRI plus cetuximab (first line); FOLFOX plus cetuximab (second line); irinotecan plus cetuximab (third line) in case of RAS/BRAF WT at each time point of progression. If at progression after the first line, the liquid biopsy assessment indicates RAS and or BRAF mutant status, patients will be treated with FOLFOX plus bevacizumab as the second line of therapy. If at progression after the second line, the liquid biopsy assessment indicates RAS and or BRAF mutant status, patients will be treated with regorafenib or trifluridine-tipiracil (investigator's choice), as third line of therapy. Each treatment will be administered using standard doses and schedules until progression of disease or unacceptable toxicity.

This study will also evaluate the activity and efficacy of cetuximab re-introduction in combination with irinotecan as third line therapy in the concept of re-challenge for those patients that will be treated in second line with FOLFOX plus bevacizumab, having a RAS or BRAF mutant disease at the time of progression after FOLFIRI plus cetuximab first line treatment. A novel characteristic of this program is that the therapeutic algorithm will be defined at each treatment decision (first line, second line and third line) in a prospective fashion in each patient by liquid biopsy assessment of RAS/BRAF status

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diagnosis of colorectal adenocarcinoma
2. Diagnosis of metastatic disease
3. RAS and BRAF wild-type status of FFPE analysis of primary colorectal cancer and/or related metastasis
4. Measurable disease according to Response Evaluation Criteria in Solid Tumors RECIST criteria, vers.1.1)
5. Male or female patients ≥ 18 years of age
6. ECOG Performance Status 0,1
7. Adequate bone marrow, liver and renal function assessed within 14 days before starting study treatment as defined by the following parameters:

   Bone marrow:
   * Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin (Hgb) ≥ 9 g/dL
   * Platelets ≥ 100 x 109/L

   Liver function:

   • Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and ALT (SGPT) ≤ 2.5 x ULN, except in patients with tumor involvement of the liver who must have AST and ALT ≤ 5 x ULN

   Renal function:

   • Serum creatinine ≤ 1.5 x ULN or 24-hour clearance ≥ 50 mL/min
8. If female and of childbearing potential, have a negative result on a pregnancy test performed a maximum of 7 days before initiation of study treatment
9. If female and of childbearing potential, or if male, agreement to use adequate contraception (e.g., abstinence, intrauterine device, oral contraceptive, or double-barrier method), during the study and until at least 3 months after last dose of study treatment administration, based on the judgment of the Investigator or a designated associate
10. Signed informed consent obtained before screening.

Exclusion Criteria:

1. Any contraindication to the use of cetuximab, Irinotecan, 5-FU, oxaliplatin, folinic acid,bevacizumab, trifluridine-tipiracil, regorafenib
2. Active uncontrolled infections, active disseminated intravascular coagulation or history of interstitial lung disease
3. Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin cancer or in situ carcinoma of the cervix
4. Pregnancy (exclusion to be ascertained by a beta hCG test)
5. Breastfeeding
6. Fertile women (<2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception•
7. Myocardial infarction, unstable angina pectoris, balloon angioplasty (PTCA) with or without stenting within the past 12 months before inclusion in the study, Grade III or IV heart failure (NYHA classification)
8. Cardiac arrhythmias requiring anti-arrhythmic therapy, with the exception of beta blockers or digoxin
9. Medical or psychological impairments associated with restricted ability to give consent or not allowing conduct of the study
10. Previous chemotherapy for the colorectal cancer with the exception of adjuvant treatment, completed at least 6 months before entering the study
11. Participation in a clinical study or experimental drug treatment within 30 days prior to study inclusion or during participation in the study
12. Known or clinically suspected brain metastases
13. History of acute or subacute intestinal occlusion or chronic inflammatory bowel disease or chronic diarrhoea
14. Severe, non-healing wounds, ulcers or bone fractures
15. Uncontrolled hypertension
16. Marked proteinuria (nephrotic syndrome)
17. Known DPD deficiency (specific screening not required)
18. Known history of alcohol or drug abuse
19. A significant concomitant disease which, in the investigating physician's opinion, rules out the patient's participation in the study
20. Absent or restricted legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
RR | up to 59 months
  Response rate (RR) for each line of treatment according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in patients with RAS/BRAF wild type (WT) mCRCregimen over 3 treatment lines in patients with RAS/BRAF wild type (WT) mCRC at start of first line therapy

SECONDARY OUTCOMES:
PFS | from 8 weeks to 59 months (from the start of therapy until the first observation of disease progression or death due to any cause)
  Progression free survival (PFS) for each line
OS | up to 59 months
  Overall Survival
AE | from screening up to 59 months
  Safety: Adverse events graded according NCI CTCAE v 5.0
EORTC Core Quality of Life questionnaire EORTC QLQ C30 | At screening, for each line of therapy at Week 4, at Week 25 of treatment start and at progression
  The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) is designed to measure cancer patients' physical, psychological and social functions. The questionnaire is composed of multi-item scales and single items
DERMATOLOGY LIFE QUALITY INDEX (DLQI) | at screening, for each line of therapy at Week 4, at Week 25 of treatment start and at progression
  The DLQI consists of 10 questions concerning patients' perception of the impact of skin diseases on different aspects of their health-related quality of life over the last week.

OTHER OUTCOMES:
Explorative objective: RR for each line of therapy | from screening up to 23 months
  the response rates for each line of therapy of RAS/BRAF WT mCRC patients who will be treated in a continuum of care strategy with cetuximab across all three therapy lines
Exploratory objective: cumulative PFS | from screening up to 23 months
  the cumulative progression free survivals of RAS/BRAF WT mCRC patients who will be treated in a continuum of care strategy with cetuximab across all three therapy lines
Explorative objective: overall survival | from screening up to 23 months
  overall survival of RAS/BRAF WT mCRC patients who will be treated in a continuum of care strategy with cetuximab across all three therapy lines
Translational analyses using next generation sequencing (NGS) technologies | At day 1 of each line of therapy
  Molecular profiles of tumor tissue and liquid biopsy samples (somatic mutations identified in tumor tissue by next generation sequencing) and surrogate markers of treatment activity (changes in molecular profile of liquid biopsies). Translational analyses of tumor biomarkers will be performed
  These include mutation in RAS, BRAF, PI3KCA; amplification of HER2, MET and loss of PTEN expression, all of which are implicated in resistance to anti-EGFR treatment.
  Moreover, 324 genes NGS panels will provide information regarding potential predictive and prognostic biomarkers of colorectal cancer disease.
  Fecal samples will be used for gut microbioma analysis, to understand how the composition of gut microbiome could influence treatment outcome and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Fortunato Ciardiello, Principal Investigator — A.O.U. dell'Università degli studi della Campania "Luigi Vanvitelli"
Locations (25):
- Italy (25):
  - A.O.U. Ospedali Riuniti, Ancona, AN
  - Ente Ecclesiastico Ospedale Generale Regionale 'F. Miulli', Acquaviva delle Fonti, BA
  - IRCCS Istituto Tumori 'Giovanni Paolo II', Bari, BA
  - Ospedale IRCCS 'Saverio de Bellis', Castellana Grotte, BA
  - Ospedale Sacro Cuore di Gesù - FATEBENEFRATELLI, Benevento, BN
  - P.O. Antonio Perrino, Brindisi, BR
  - A.O.U. Cagliari - Presidio Policlinico D. Casula, Monserrato, CA
  - A.R.N.A.S. Garibaldi - P.O. Garibaldi-Nesima, Catania, CT
  - A.O.U. Mater Domini, Catanzaro, CZ
  - Fondazione IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, FG
  - P.O. 'Vito Fazzi', Lecce, LE
  - A.O. 'Pia Fondazione Cardinale G. Panico', Tricase, LE
  - Istituto Europeo di Oncologia, Milan, MI
  - A.O.U. Policlinico 'P. Giaccone', Palermo, PA
  - Istituto Oncologico Veneto IRCCS, Padua, PD
  - A.O.U. Pisana, Pisa, PI
  - A.O. San Carlo, Potenza, PZ
  - A.U.S.L. - IRCCS di Reggio Emilia - P.O. Arcispedale S.Maria Nuova, Reggio Emilia, RE
  - A.S.P. Ragusa - Ospedale Maria Paternò Arezzo, Ragusa, RG
  - A.O. San Camillo-Forlanini, Roma, RM
  - Fondazione Policlinico Universitario 'Agostino Gemelli' IRCCS, Roma, RM
  - Ospedale San Giuseppe Moscati, Statte, TA
  - A.O. Ordine Mauriziano, Torino, TO
  - A.O.U. dell'Università degli studi della Campania "Luigi Vanvitelli", Napoli
  - Istituto Nazionale Tumori 'Fondazione G. Pascale', Napoli

REFERENCES:
- [Derived] Martini G, Ciardiello D, Napolitano S, Martinelli E, Troiani T, Latiano TP, Avallone A, Normanno N, Di Maio M, Maiello E, Ciardiello F. Efficacy and safety of a biomarker-driven cetuximab-based treatment regimen over 3 treatment lines in mCRC patients with RAS/BRAF wild type tumors at start of first line: The CAPRI 2 GOIM trial. Front Oncol. 2023 Feb 13;13:1069370. doi: 10.3389/fonc.2023.1069370. eCollection 2023. PMID 36860319